CLINICAL TRIAL: NCT04084067
Title: Indocyanine Green (ICG) Guided Tumor Resection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICGLOW; NCI-2019-06146 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Neoplastic Disease; Solid Tumor
Keywords: Ewing Sarcoma; Liver tumor; Lymphoma; Metastatic pulmonary deposits; Neoplastic Disease; Neuroblastoma; Non-Rhabdomyosarcoma Soft Tissue Sarcoma; Nodules of unknown etiology; Osteosarcoma; Solid Tumor; Rhabdomyosarcoma; Renal tumors; Rare tumors
MeSH Terms: conditions — Neoplasms; Sarcoma, Ewing; Carcinoma, Hepatocellular; Lymphoma; Neuroblastoma; Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Carcinoma, Renal Cell | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Indocyanine green (ICG) (Experimental): Participants will receive a single dose of 1.5 mg/kg of ICG intravenously over 15 minutes prior to surgery.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — IV
  Other Names: IC-GREEN™; ICG

SUMMARY:
This is a study to assess the ability of Indocyanine Green (ICG) to identify neoplastic disease. For many pediatric solid tumors, complete resection of the primary site and/or metastatic deposits is critical for achieving a cure. An optimal intra-operative tool to help visualize tumor and its margins would be of benefit. ICG real-time fluorescence imaging is a technique being used increasingly in adults for this purpose. We propose to use it during surgery for pediatric malignancies. All patients with tumors that require localization for resection or biopsy of the tumor and/or metastatic lesions will be eligible.

Primary Objective

To assess the feasibility of Indocyanine Green (ICG)-mediated near-infrared (NIR) imagery to identify neoplastic disease during the conduct of surgery to resect neoplastic lesions in children and adolescents. NIR imaging will be done at the start of surgery to assess NIR-positivity of the lesion(s) and at the end of surgery to assess completeness of resection. Separate assessments will be made for the following different histologic categories:

1. Osteosarcoma
2. Neuroblastoma
3. Metastatic pulmonary deposits - closed to accrual

Exploratory Objectives

1. To compare the ICG uptake by primary vs metastatic site and pre-treated (chemotherapy, radiation, or both) vs non-pre-treated.
2. Assess the sensitivity and specificity of NIR imagery to find additional lesions not identified by standard of care intraoperative inspection and tactile feedback.
3. Assess the sensitivity and specificity of NIR imagery to find additional lesions not identified on preoperative diagnostic imaging.
4. Assess the sensitivity and specificity of NIR imagery for identifying residual disease at the conclusion of a tumor resection.

Separate assessments will be made for the following different histologic categories based on their actual enrollment; this includes but is not limited to analyzing multiple arms together:

1. Ewing Sarcoma
2. Rhabdomyosarcoma (RMS)
3. Non-Rhabdomyosarcoma Soft Tissue Sarcoma (NRSTS)
4. Renal tumors
5. Liver tumors, lymphoma, other rare tumors, and nodules of unknown etiology

DETAILED DESCRIPTION:
This trial is a single center open-label study. Patients with a solid tumor or lymphoma who require resection either for therapeutic or diagnostic intent will be included.

Indocyanine Green (ICG) is an FDA-approved drug. Prior to surgery, patients will receive a single dose of ICG intravenously.

During surgery, after the surgeon identifies the mass through visual (seen with the naked eye) and or tactile methods (palpated), the patient will have his/her tumor field imaged by Iridium system optimized for detection of ICG (EleVision™ IR Platform). The entire procedure will be photo- documented and recorded.

The EleVision™ system records images in real time, calculates percentages, and captures the data. At least three different areas of the tumor will be measured. If the tumor cannot be identified by visual inspection or palpation, NIR-imaging will be used in an attempt to locate the lesion. The surrounding area will be inspected and measured to screen for additional sites of metastatic disease. After tumor resection, residual fluorescence in the surgical resection bed will be measured.

Direct subject participation in the trial will last for the period of time from injection of the ICG the day before surgery and until 24 hours post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary or relapsed solid tumor or lymphoma who require excision of the tumor or metastatic lesions.

Exclusion Criteria:

* Subjects with a history of iodide allergies.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Patients with benign pathology.
* Patients with brain tumors.
* Pregnant female.
* Patients with unilateral Wilms Tumor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity rates of the ICG guided neoplastic disease identification | up to 24 hours post-surgery
  Participants in each of the primary objective categories will be evaluated for this objective.

OTHER OUTCOMES:
Sensitivity rates of the ICG guided neoplastic disease identification | up to 24 hours post-surgery
  Participants in each of the exploratory objective categories will be evaluated for this objective.
Sensitivity and specificity rates of the ICG guided residual (lymph node and tumor bed) neoplastic disease identification | up to 24 hours post-surgery
  Participants in each of the primary and exploratory objective categories will be evaluated for this objective.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Talbot, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- [Derived] Abdelhafeez AH, Mothi SS, Pio L, Mori M, Santiago TC, McCarville MB, Kaste SC, Pappo AS, Talbot LJ, Murphy AJ, Davidoff AM. Feasibility of indocyanine green-guided localization of pulmonary nodules in children with solid tumors. Pediatr Blood Cancer. 2023 Oct;70(10):e30437. doi: 10.1002/pbc.30437. Epub 2023 May 17. PMID 37194488
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols